CLINICAL TRIAL: NCT03319043
Title: Observation of the Respiratory Impedance and Inflammation in Cough Variant Asthma Patients Treated in Combination of Chanqin Granules.
Brief Title: Observation of Cough Variant Asthma Treated in Combination of Chanqin Granules.
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20164Y0199
Record Dates: First submitted 2017-08-20; First posted 2017-10-24 (Actual); Last update posted 2017-10-24 (Actual); Status verified 2016-12

CONDITIONS: Cough Variant Asthma
Keywords: Cough Variant Asthma; impedance; inflammation; Chanqin granules
MeSH Terms: conditions — Cough-Variant Asthma; Inflammation | interventions — Budesonide; Formoterol Fumarate

STUDY DESIGN:
Intervention Model Description: A total of 120 eligible participants will be randomly allocated to the placebo group and treatment group in a 1:1 ratio. Randomized sequences of each center and every packed drug were generated by an independent professor at the Drug Clinical Research Center of Shanghai University of TCM, using a stratified block randomization method with 30 blocks of block size 8 based on the PROC PLAN function of the SAS 9.2 software analysis system (SAS Institute, Cary, NC, USA).
Who Masked: Participant, Care Provider, Investigator
Masking Description: Randomization sequences will be concealed in lightproof, sealed envelopes kept by a specified project manager and the sponsor, who are not involved in the recruitment, intervention, assessment, or statistical analysis. The treatment allocation will be blinded to the participants and investigators throughout the study, and the outcome assessors and statisticians will not be involved in the participants' screening and allocation. Each patient will receive a unique randomized number corresponding to the drug according to the group allocation. Furthermore, the intervention group type will be replaced by the letter A, B as blind codes of allocation. The blind codes will not be disclosed until the statistical analysis is completed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- treatment group (Experimental): patients are treated with Budesonide + Formoterol Fumarate dry powder (160/4.5ug bid) for inhalation and additional Chanqin granules 10g three times a day. All granules will be taken orally with 200 ml warm water.
  Interventions: Drug: Chanqin granules
- controlled group (Placebo Comparator): patients enrolled in the research are treated with Budesonide + Formoterol Fumarate dry powder (160/4.5ug bid) for inhalation and Chanqin analogous granules. All granules will be taken orally with 200 ml warm water.
  Interventions: Drug: Chanqin granules

INTERVENTIONS:
Drug: Chanqin granules — All patients enrolled in the research are treated with Budesonide + Formoterol Fumarate dry powder (160/4.5ug bid) for inhalation. Patients in treatment group are given additional Chanqin granules 10g three times a day; and analogous for the controlled group.
  Other Names: Budesonide + Formoterol Fumarate; Chanqin granules analogous

SUMMARY:
This single-center, randomized, double-blind, placebo-controlled trial was undertaken at an outpatient clinic in Shuguang Hospital. Newly diagnosed cough variant asthma adult patients with the T.C.M. pattern of pathogenic-wind are randomly divided into treatment and control group, with 60 patients in each group. Clinical observation of the Respiratory Impedance and Inflammation in Cough Variant Asthma adults reated in Combination of Chanqin Granules.

DETAILED DESCRIPTION:
This single-center, randomized, double-blind, placebo-controlled trial was undertaken at an outpatient clinic in Shuguang Hospital. Newly diagnosed cough variant asthma adult patients with the T.C.M. pattern of pathogenic-wind are randomly divided into treatment and control group, with 60 patients in each group. All patients enrolled are treated with Budesonide + Formoterol Fumarate dry power (160/4.5ug bid) for inhalation. The treatment group are given additional Chanqin granulate (10g bid) and placebo granulate for controlled group. Investigators hypothesis that Chanqin granules may reduce day & night cough score as well as the respiratory impedance, inflammation statues, and improve T.C.M. syndrome after 8 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of cough variant asthma according to Western medicine
2. Diagnosis of cough with pathogenic wind syndrome according to TCM
3. Aged between 18 to 70 years, regardless of gender, race or educational and economic status
4. The cough symptom should last for at least 8 weeks

4. Willingness to participate and to sign the informed consent form

Exclusion Criteria:

1. Patients with history of smoking (or quite smoking for less than 6 months)
2. Systemic use of corticosteroids in the past 4 weeks
3. Upper or lower respiratory tract infection in the past 4 weeks
4. Incapable of corporation with spirometry and FeNO test
5. Other chronic respiratory disease eg: COPD, pulmonary cirrhosis
6. Women who are pregnant or preparing to become pregnant or breast feeding women

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2017-11-01 (Estimated); Primary Completion 2018-12-30 (Estimated); Study Completion 2019-06-30 (Estimated)

PRIMARY OUTCOMES:
Impulse Oscillometry | 2 week
  The patients will be seated comfortably in a nonswivel chair. Nose clips were applied and a special mouthpiece will be used. For Impulse Oscillometry measurements (MasterScreen, CareFusion, San Diego, California) are performed according to the protocols of the European Respiratory Society. Patients will be advised to cradle their cheeks with their hands. Patients are allowed to breathe normally while the loudspeaker delivere intermittent multi-frequency impulses over a minimum of a 30-s period. A trained technician will guide and assist the patient during the procedure, which involved three to five sinusoidal readings, depending on the incidence of cough, swallowing, and holding of breath. The recordings with the best coherence at frequencies from 5 to 30 Hz will be chosen. The technician is also trained to capture subclinical leaks through the mouthpiece, and leaky recordings will be discarded. The Impulse Oscillometry parameters measured are Zrs、R5、R20、X5.

SECONDARY OUTCOMES:
Cough severity | 2 week
  Cough severity is measured by a validated verbal category-descriptive (VCD) scores which patients reported. =The scale has 6 discrete values: 0=no cough; 1=one short period of mild cough without hardship; 2=some short periods of cough without much hardship; 3=frequent coughing that does not affect normal daily life or sleep; 4=serious coughing that is very frequent and interferes with normal daily life or sleep; 5=distressing continuous coughing that did not stop for 24 h.
Exhaled nitric oxide | 2 week
  Exhaled nitric oxide is measured using a portable analyzer, the NIOX MINO (Aerocrine AB, Solna, Sweden). Participants performe a 10 seconds slow steady exhalation. Three successive recordings at 1-minute intervals, expressed as parts per billion (ppb), are made.

CONTACTS AND LOCATIONS:
Overall Officials: XUAN CHEN, Master, Study Director — Shanghai University of T.C.M.
Locations (1):
- Shuguang Hospital affiliated to Shanghai University of Traditional Chinese Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
Access to these data and associated recommendations generated under the project will be available for educational, research and non-profit purposes.

REFERENCES:
- [Background] Saadeh C, Saadeh C, Cross B, Gaylor M, Griffith M. Advantage of impulse oscillometry over spirometry to diagnose chronic obstructive pulmonary disease and monitor pulmonary responses to bronchodilators: An observational study. SAGE Open Med. 2015 Apr 6;3:2050312115578957. doi: 10.1177/2050312115578957. eCollection 2015. PMID 26770777
- [Background] Shimoda T, Obase Y, Kishikawa R, Iwanaga T, Miyatake A, Kasayama S. The fractional exhaled nitric oxide and serum high sensitivity C-reactive protein levels in cough variant asthma and typical bronchial asthma. Allergol Int. 2013 Jun;62(2):251-7. doi: 10.2332/allergolint.12-OA-0515. Epub 2013 Apr 25. PMID 23612495
- [Background] Bickel S, Popler J, Lesnick B, Eid N. Impulse oscillometry: interpretation and practical applications. Chest. 2014 Sep;146(3):841-847. doi: 10.1378/chest.13-1875. PMID 25180727
- [Result] Berry MA, Shaw DE, Green RH, Brightling CE, Wardlaw AJ, Pavord ID. The use of exhaled nitric oxide concentration to identify eosinophilic airway inflammation: an observational study in adults with asthma. Clin Exp Allergy. 2005 Sep;35(9):1175-9. doi: 10.1111/j.1365-2222.2005.02314.x. PMID 16164444